CLINICAL TRIAL: NCT04086992
Title: Decreasing Parental Stress and Costs While Improving Overall Satisfaction of Caregivers of Infants With Infantile Spasms on ACTH Therapy Utilizing Innovative Telemedicine Technology: A Randomized Study
Brief Title: Decreasing Parental Stress of Caregivers of Infants With Infantile Spasms by Using Telemedicine Technology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Colorado, Denver (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-0579
Record Dates: First submitted 2019-08-27; First posted 2019-09-12 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Infantile Spasms, Non-Intractable
Keywords: Infantile Spasms; parental stress; ACTH; remote monitoring
MeSH Terms: conditions — Spasms, Infantile | interventions — Remote Patient Monitoring

STUDY DESIGN:
Intervention Model Description: Patients with infantile spasms will be randomized into either the control group that will receive traditional follow-up or the intervention group that will receive remote monitoring for follow-up. Both groups will complete surveys to collect data on parental stress, direct and indirect costs, and overall satisfaction with therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): This group will continue to receive standard care for ACTH monitoring and follow-up with includes blood pressure by the patient's PCP while on therapy, a one week nursing follow-up phone call, and a two-week EEG and Neurology appointment.
- Intervention Group (Experimental): This group will be provided remote monitoring technology where they will be able to monitor blood pressure at home. In addition, they will receive a nurse-led telemedicine visit at one week and three weeks of therapy. Like the control group, they will still receive a two-week EEG and Neurology appointment.
  Interventions: Other: Remote monitoring

INTERVENTIONS:
Other: Remote monitoring — Caregivers will be able to monitor blood pressure from home and upload in a cloud-based application on a hand-held tablet. In addition, this technology will administer surveys to the caregiver to assess for therapy side effects and adherence. Nurse-led telemedicine visits will also be utilized. The healthcare team will be able to monitor these parameters remotely.
  Arms: Intervention Group

SUMMARY:
This study plans to learn more about how the use of new telemedicine technology can help with parental stress, costs, and overall satisfaction in care. Investigators are studying this in families who have children with a specific seizure type called infantile spasms and being treated with a medication called ACTH (adrenocorticotropic hormone). Infantile spasms is a rare epileptic encephalopathy that occurs within the first two years of life. It is associated with complicated and expensive treatment and poor developmental outcomes. Participants will be randomly placed in one of two groups. The first group will continue with the traditional monitoring practices primarily performed by their pediatrician. The second group will use telemedicine technology to be monitored. Investigators will then compare the two groups to see if there are any differences in parental stress, costs of care, and/or overall satisfaction with care.

The primary hypothesis is that compared to those utilizing usual monitoring, parents/caregivers of infants with IS treated with ACTH utilizing nurse-led remote biometric monitoring will report less parenting stress at 2 and 4 weeks of treatment.

DETAILED DESCRIPTION:
Infantile Spasms, historically call West Syndrome, is an infantile epileptic encephalopathy, typically occurring within the first two years of life. Infantile Spasms is often characterized by hypsarrhythmia on encephalogram (EEG) and developmental plateau or regression. It is estimated that Infantile Spasms affects 2 to 5 per 10,000 live births. The etiology of Infantile Spasms is varied and often unclear at the time of diagnosis. In almost half of cases it is linked to hypoxic-ischemic encephalopathy, chromosomal abnormalities, perinatal stroke, tuberous sclerosis complex, or periventricular leukomalacia or hemorrhage.

While historically treatment options have been widely variable, over the past several years three pharmacologic therapies have been adopted, including ACTH, oral corticosteroids (OCS), and vigabatrin.

ACTH was approved for use for multiple neurologic conditions in 1952 and specifically for Infantile Spasms in 2010. Unfortunately, as a hormone therapy, ACTH carries several potentially severe side effects including adrenal insufficiency, immunosuppression, electrolyte imbalances, and more commonly elevated blood pressure thought to lead to serious cardiac changes.

Complexity of ACTH therapy requires close monitoring. ACTH is administered intramuscularly twice a day for the initial two weeks with a complicated weaning schedule over the subsequent 2 weeks. Between the required monitoring and complicated administration regimen, ACTH therapy is often overwhelming and confusing for caregivers, and can lead to medication errors.

Unfortunately, primary care (PCP) monitoring for ACTH has proved to be inconsistent. Barriers for families have included: families without an identified PCP, families without the means to get to their PCP at the recommended intervals (rural location or inadequate transportation), PCP's without the correct equipment to monitor infants, limited office hours, and PCP with little comfort in managing side-effects when they present. This has resulted in disjointed care, and last-minute attempts to obtain needed monitoring in less-than-ideal settings (e.g., urgent care, hospital, neurology clinic) - all with additional expense to families.

Treatment with ACTH is associated with high direct and indirect costs. Treatment of Infantile Spasms with ACTH carries a significant financial burden for families. In August 2007, the cost for one vial of ACTH, then manufactured by Questcor Pharmaceuticals and now by Mallinckrodt Pharmaceuticals, increased from $1650 to $23,000. Current, non-discounted pricing is $34,400 per vial. The average therapy calls for 3-4 vials, with a total price tag between $103,200 and $137,600. Any potential for medication error further exacerbates costs of therapy.

Consumer-incurred costs of ACTH therapy have not previously been reported. Direct costs of ACTH therapy for caregivers include, at a minimum, the out-of-pocket expense for the drug as well as required PCP, neurology, and EEG follow-up. It is not uncommon, due to complications of monitoring, that caregivers sustain additional direct costs seeking monitoring in unplanned ways (e.g., urgent care/ED visits). In addition, prophylactic treatment with antibiotics and H2 blockers to combat potential side effects is necessary and adds to caregiver expense. Indirect costs include loss of productivity due to work absences and non-paid loss of productivity (e.g., homemaker). Expense of transportation and travel can also be significant.

Considering the potential severe side-effects of ACTH, the complicated medication regime, the rigorous required follow-up, the costs inherent in the therapy alone and those due to complications, it is hypothesized that parenting stress for parents of babies with IS is high. Support for these families is critical to successful ACTH therapy. Historically at Children's Hospital Colorado, there has been no structured support outside of the initial admission for diagnosis/start of therapy and follow-up neurology appointments. This study is intended to explore and compare parenting stress of parents/caregivers caring for babies with IS being treated with ACTH and secondarily, overall treatment satisfaction.

Remote biometric monitoring led by highly skilled registered nurses could offer a novel, feasible, cost-effective strategy to support families of infants with IS during treatment with ACTH. Although there is currently no published literature exploring the use of telehealth or remote monitoring in the specific treatment of Infantile Spasms, its successful use in other complex conditions underscores its potential for benefit. In addition to optimization of disease-related outcomes, remote monitoring has high potential to reduce financial burden and parenting stress on parent/caregivers.

This proposed study will utilize a prospective randomized clinical trial design. - Infants and caregivers of infants who meet the inclusion criteria will be invited to participate. They will be randomized to the intervention or usual care group in accordance with a random number generator program through the Biostatistics Core at CHCO. Randomization will be stratified by payor source.

The study hypotheses include:

1. Compared to those utilizing usual monitoring, parents/caregivers of infants with IS treated with ACTH utilizing nurse-led remote biometric monitoring will report less parenting stress at 2 and 4 weeks of treatment.
2. Compared to those utilizing usual monitoring, parents/caregivers of infants with IS treated with 4 weeks of ACTH utilizing nurse-led remote biometric monitoring will experience a decrease in direct (including travel) and indirect cost of care.
3. Compared to those utilizing usual monitoring, parents/caregivers of infants with IS treated with ACTH utilizing nurse-led remote biometric monitoring will experience greater overall satisfaction with treatment.

All caregivers will be given the standard education on Infantile Spasms, ACTH and ACTH administration.

The control group will continue to receive standard care for ACTH monitoring and follow-up, which includes:

1. Blood pressure monitoring by PCP recommended to occur a minimum of two times per week. Depending on the results and PCP's comfort in managing any aberrant results, the PCP may or may not share them with the patient's primary neurologist.
2. Nurse follow-up phone call at 1 week of therapy to assess spasm frequency, monitoring and medication adherence, side-effects, complications of therapy, validate the dosing schedule, confirm required follow-up appointments (Neurology and EEG), answer any questions, and provide support. Data collected during these calls is routed to the patient's primary neurologist for review.
3. EEG follow-up at 2 weeks of therapy - results are sent to primary neurologist.
4. Neurology appointment at 2 weeks of therapy

The intervention group will receive and be instructed on the use of a re-useable digital health kit that will include an electronic tablet with integrated monitoring and telehealth software and manual or automatic blood pressure machine with appropriate sized cuff. The software utilized is web-based and has the capability to integrate into an organization's electronic health record. It allows for the real-time monitoring by healthcare professionals and the establishment of alerts. Appropriate research personnel will be responsible for this monitoring. In addition to biometric monitoring, the software allows for individualized health and other surveys to gain immediate patient feedback. Finally, the tablet and software support video telemedicine visits in the patient home.

The following interventions will be utilized in the intervention group:

1. Caregivers will take blood pressure three times per week (ideally, Monday, Wednesday, Friday) and will uploaded into the monitoring software/tablet. A neurology nurse will monitor these results, transcribe them into the patient's medical record, and route them to the patient's primary neurologist for review and potential follow-up.
2. Caregivers will complete a twice-a-week side-effect and adherence survey in the software/tablet. The results of this survey will be transcribed into the patient's medical record and routed to the patient's primary neurologist for review and potential follow-up.
3. A neurology nurse will conduct a video telehealth visit with the caregiver to assess spasm frequency, monitoring and medication adherence, side-effects, complications of therapy, validate the dosing schedule, confirm required follow-up appointments (Neurology and EEG), answer any questions, and provide support between days 7-10 and again between days 21-24 of therapy. This will be documented as a telehealth nurse-visit and routed to the patient's primary neurologist for review and potential follow-up.
4. EEG follow-up at 2 weeks of therapy - results are sent to primary neurologist.
5. Neurology appointment at 2 weeks of therapy

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to CHCO, Anschutz and Colorado Springs hospitals, under the age of 30 months with a primary diagnosis of Infantile Spasms and started on first-time ACTH and their primary caregiver (parent/guardian).

Exclusion Criteria:

* Infants with recurrent Infantile Spasms and retreatment with ACTH and their primary caregiver (parent/guardian).
* Infants with existing home health nursing services and their primary caregiver (parent/guardian).
* Infants with prolonged inpatient admissions beyond 7 days after initiation on ACTH and their primary caregiver (parent/guardian).
* Infants whose caregivers do not read, write, and/or speak English with sufficient proficiency to provide informed consent and their primary caregiver (parent/guardian).
* Neonates less than 31 days old and their primary caregiver (parent/guardian).
* Infants that have been hospitalized since birth and their primary caregiver (parent/guardian).
* Infants that are wards of the state and their primary caregiver (guardian).
* Infants that reside in a geographic location with no major network cell service and their primary caregiver (parent/guardian).

Ages: 31 Days to 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Compare parental stress between intervention group and control group | At study enrollment (prior to hospital discharge)
  Parental stress will be measures by the Pediatric Inventory for Parents (PIP), a previously validated survey. The PIP is scored separately for each of the 4 domains (Communication, Emotional Distress, Medical Care, Role Function), across 2 scales: Frequency (F) and Difficulty (D). The range for each of the scales is 42-210, with a higher score on either scale indicating more stress.
Compare parental stress between intervention group and control group | Mid-therapy (between week 2 and 3 of therapy)
  Parental stress will be measures by the Pediatric Inventory for Parents (PIP), a previously validated survey. The PIP is scored separately for each of the 4 domains (Communication, Emotional Distress, Medical Care, Role Function), across 2 scales: Frequency (F) and Difficulty (D). The range for each of the scales is 42-210, with a higher score on either scale indicating more stress.
Compare parental stress between intervention group and control group | At therapy completion (end of week 4, with 7 days to complete)
  Parental stress will be measures by the Pediatric Inventory for Parents (PIP), a previously validated survey. The PIP is scored separately for each of the 4 domains (Communication, Emotional Distress, Medical Care, Role Function), across 2 scales: Frequency (F) and Difficulty (D). The range for each of the scales is 42-210, with a higher score on either scale indicating more stress.
Compare overall satisfaction with treatment between intervention group and control group | At therapy completion (end of week 4, with 7 days to complete)
  Overall treatment satisfaction will be measured by the Treatment Satisfaction Questionnaire for Medications, version 9 (TSQM v9) survey. This is a previously validated survey. The scores for the TSQM v9 can range from 1-100, with a higher score indicating greater satisfaction.
Compare expenses between intervention group and control group | At mid-therapy (between week 2 and 3 of therapy)
  Caregivers will be asked to provide details on both direct and indirect costs incurred during therapy. This will be measured by collecting both healthcare utilizations rates, actual out-of-pocket expenses, and lost productivity measures. Combined direct and indirect expenses will be combined and compared.
Compare expenses between intervention group and control group | At therapy completion (end of week 4, with 7 days to complete)
  Caregivers will be asked to provide details on both direct and indirect costs incurred during therapy. This will be measured by collecting both healthcare utilizations rates, actual out-of-pocket expenses, and lost productivity measures. Combined direct and indirect expenses will be combined and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer D Coffman, BSN, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.

REFERENCES:
- [Background] Knupp KG, Coryell J, Nickels KC, Ryan N, Leister E, Loddenkemper T, Grinspan Z, Hartman AL, Kossoff EH, Gaillard WD, Mytinger JR, Joshi S, Shellhaas RA, Sullivan J, Dlugos D, Hamikawa L, Berg AT, Millichap J, Nordli DR Jr, Wirrell E; Pediatric Epilepsy Research Consortium. Response to treatment in a prospective national infantile spasms cohort. Ann Neurol. 2016 Mar;79(3):475-84. doi: 10.1002/ana.24594. Epub 2016 Feb 13. PMID 26704170
- [Background] Osborne JP, Lux AL, Edwards SW, Hancock E, Johnson AL, Kennedy CR, Newton RW, Verity CM, O'Callaghan FJ. The underlying etiology of infantile spasms (West syndrome): information from the United Kingdom Infantile Spasms Study (UKISS) on contemporary causes and their classification. Epilepsia. 2010 Oct;51(10):2168-74. doi: 10.1111/j.1528-1167.2010.02695.x. Epub 2010 Aug 17. PMID 20726878
- [Background] Iype M, Saradakutty G, Kunju PA, Mohan D, Nair MK, George B, Ahamed SM. Infantile spasms: A prognostic evaluation. Ann Indian Acad Neurol. 2016 Apr-Jun;19(2):228-35. doi: 10.4103/0972-2327.173314. PMID 27293335
- [Background] Widjaja E, Go C, McCoy B, Snead OC. Neurodevelopmental outcome of infantile spasms: A systematic review and meta-analysis. Epilepsy Res. 2015 Jan;109:155-62. doi: 10.1016/j.eplepsyres.2014.11.012. Epub 2014 Nov 22. PMID 25524855
- [Background] Kossoff EH, Hartman AL, Rubenstein JE, Vining EP. High-dose oral prednisolone for infantile spasms: an effective and less expensive alternative to ACTH. Epilepsy Behav. 2009 Apr;14(4):674-6. doi: 10.1016/j.yebeh.2009.01.023. Epub 2009 Feb 4. PMID 19435579
- [Background] Lux AL, Edwards SW, Hancock E, Johnson AL, Kennedy CR, Newton RW, O'Callaghan FJ, Verity CM, Osborne JP; United Kingdom Infantile Spasms Study. The United Kingdom Infantile Spasms Study (UKISS) comparing hormone treatment with vigabatrin on developmental and epilepsy outcomes to age 14 months: a multicentre randomised trial. Lancet Neurol. 2005 Nov;4(11):712-7. doi: 10.1016/S1474-4422(05)70199-X. PMID 16239177
- [Background] Go CY, Mackay MT, Weiss SK, Stephens D, Adams-Webber T, Ashwal S, Snead OC 3rd; Child Neurology Society; American Academy of Neurology. Evidence-based guideline update: medical treatment of infantile spasms [RETIRED]. Report of the Guideline Development Subcommittee of the American Academy of Neurology and the Practice Committee of the Child Neurology Society. Neurology. 2012 Jun 12;78(24):1974-80. doi: 10.1212/WNL.0b013e318259e2cf. PMID 22689735
- [Background] Wray CD, Benke TA. Effect of price increase of adrenocorticotropic hormone on treatment practices of infantile spasms. Pediatr Neurol. 2010 Sep;43(3):163-6. doi: 10.1016/j.pediatrneurol.2010.04.005. PMID 20691936
- [Background] Ibrahim A, Umar UI, Usman UM, Owolabi LF. Economic evaluation of childhood epilepsy in a resource-challenged setting: A preliminary survey. Epilepsy Behav. 2017 Nov;76:84-88. doi: 10.1016/j.yebeh.2017.08.023. Epub 2017 Sep 13. PMID 28917500
- [Background] Burton WN, Chen CY, Conti DJ, Pransky G, Edington DW. Caregiving for ill dependents and its association with employee health risks and productivity. J Occup Environ Med. 2004 Oct;46(10):1048-56. doi: 10.1097/01.jom.0000141830.72507.32. PMID 15602179
- [Background] Bator EX, Gleason JM, Lorenzo AJ, Kanaroglou N, Farhat WA, Bagli DJ, Koyle MA. The burden of attending a pediatric surgical clinic and family preferences toward telemedicine. J Pediatr Surg. 2015 Oct;50(10):1776-82. doi: 10.1016/j.jpedsurg.2015.06.005. Epub 2015 Jun 20. PMID 26195452
- [Background] Wirrell EC, Wood L, Hamiwka LD, Sherman EM. Parenting stress in mothers of children with intractable epilepsy. Epilepsy Behav. 2008 Jul;13(1):169-73. doi: 10.1016/j.yebeh.2008.02.011. Epub 2008 Mar 11. PMID 18337182
- [Background] Chiou HH, Hsieh LP. Parenting stress in parents of children with epilepsy and asthma. J Child Neurol. 2008 Mar;23(3):301-6. doi: 10.1177/0883073807308712. Epub 2008 Jan 8. PMID 18182646
- [Background] Modi AC. The impact of a new pediatric epilepsy diagnosis on parents: parenting stress and activity patterns. Epilepsy Behav. 2009 Jan;14(1):237-42. doi: 10.1016/j.yebeh.2008.10.009. Epub 2008 Nov 26. PMID 18977459
- [Background] Ong MK, Romano PS, Edgington S, Aronow HU, Auerbach AD, Black JT, De Marco T, Escarce JJ, Evangelista LS, Hanna B, Ganiats TG, Greenberg BH, Greenfield S, Kaplan SH, Kimchi A, Liu H, Lombardo D, Mangione CM, Sadeghi B, Sadeghi B, Sarrafzadeh M, Tong K, Fonarow GC; Better Effectiveness After Transition-Heart Failure (BEAT-HF) Research Group. Effectiveness of Remote Patient Monitoring After Discharge of Hospitalized Patients With Heart Failure: The Better Effectiveness After Transition -- Heart Failure (BEAT-HF) Randomized Clinical Trial. JAMA Intern Med. 2016 Mar;176(3):310-8. doi: 10.1001/jamainternmed.2015.7712. PMID 26857383
- [Background] McElroy I, Sareh S, Zhu A, Miranda G, Wu H, Nguyen M, Shemin R, Benharash P. Use of digital health kits to reduce readmission after cardiac surgery. J Surg Res. 2016 Jul;204(1):1-7. doi: 10.1016/j.jss.2016.04.028. Epub 2016 Apr 23. PMID 27451860
- [Background] DeAlleaume L, Parnes B, Zittleman L, Sutter C, Chavez R, Bernstein J, LeBlanc W, Dickinson M, Westfall JM. Success in the Achieving CARdiovascular Excellence in Colorado (A CARE) Home Blood Pressure Monitoring Program: A Report from the Shared Networks of Colorado Ambulatory Practices and Partners (SNOCAP). J Am Board Fam Med. 2015 Sep-Oct;28(5):548-55. doi: 10.3122/jabfm.2015.05.150024. PMID 26355126
- [Background] Siehr SL, Norris JK, Bushnell JA, Ramamoorthy C, Reddy VM, Hanley FL, Wright GE. Home monitoring program reduces interstage mortality after the modified Norwood procedure. J Thorac Cardiovasc Surg. 2014 Feb;147(2):718-23.e1. doi: 10.1016/j.jtcvs.2013.04.006. Epub 2013 May 8. PMID 23663957
- [Background] Ladapo JA, Turakhia MP, Ryan MP, Mollenkopf SA, Reynolds MR. Health Care Utilization and Expenditures Associated With Remote Monitoring in Patients With Implantable Cardiac Devices. Am J Cardiol. 2016 May 1;117(9):1455-62. doi: 10.1016/j.amjcard.2016.02.015. Epub 2016 Feb 17. PMID 26996767
- [Background] Robinson JD, Prochaska JD, Yngve DA. Pre-surgery evaluations by telephone decrease travel and cost for families of children with cerebral palsy. SAGE Open Med. 2017 Jul 23;5:2050312117720046. doi: 10.1177/2050312117720046. eCollection 2017. PMID 28839936
- [Background] Gevers M, van Genderingen HR, Lafeber HN, Hack WW. Accuracy of oscillometric blood pressure measurement in critically ill neonates with reference to the arterial pressure wave shape. Intensive Care Med. 1996 Mar;22(3):242-8. doi: 10.1007/BF01712244. PMID 8727439
- [Background] Park MK, Menard SM. Accuracy of blood pressure measurement by the Dinamap monitor in infants and children. Pediatrics. 1987 Jun;79(6):907-14. PMID 3588145
- [Background] Friesen RH, Lichtor JL. Indirect measurement of blood pressure in neonates and infants utilizing an automatic noninvasive oscillometric monitor. Anesth Analg. 1981 Oct;60(10):742-5. PMID 7197478
- [Background] Cullen PM, Dye J, Hughes DG. Clinical assessment of the neonatal Dinamap 847 during anesthesia in neonates and infants. J Clin Monit. 1987 Oct;3(4):229-34. doi: 10.1007/BF03337376. PMID 3681356
- [Background] Chia F, Ang AT, Wong TW, Tan KW, Fung KP, Lee J, Khin K. Reliability of the Dinamap non-invasive monitor in the measurement of blood pressure of ill Asian newborns. Clin Pediatr (Phila). 1990 May;29(5):262-7. doi: 10.1177/000992289002900502. PMID 2340688
- [Background] Colan SD, Fujii A, Borow KM, MacPherson D, Sanders SP. Noninvasive determination of systolic, diastolic and end-systolic blood pressure in neonates, infants and young children: comparison with central aortic pressure measurements. Am J Cardiol. 1983 Oct 1;52(7):867-70. doi: 10.1016/0002-9149(83)90430-7. PMID 6624679
- [Background] Nelson RM, Stebor AD, Groh CM, Timoney PM, Theobald KS, Friedman BA. Determination of accuracy in neonates for non-invasive blood pressure device using an improved algorithm. Blood Press Monit. 2002 Apr;7(2):123-9. doi: 10.1097/00126097-200204000-00006. PMID 12048430
- [Background] Stergiou GS, Nasothimiou E, Giovas P, Kapoyiannis A, Vazeou A. Diagnosis of hypertension in children and adolescents based on home versus ambulatory blood pressure monitoring. J Hypertens. 2008 Aug;26(8):1556-62. doi: 10.1097/HJH.0b013e328301c411. PMID 18622232
- [Background] Flynn JT, Kaelber DC, Baker-Smith CM, et al; SUBCOMMITTEE ON SCREENING AND MANAGEMENT OF HIGH BLOOD PRESSURE IN CHILDREN. Clinical Practice Guideline for Screening and Management of High Blood Pressure in Children and Adolescents. Pediatrics. 2017; 140(3):e20171904. Pediatrics. 2017 Dec;140(6):e20173035. doi: 10.1542/peds.2017-3035. No abstract available. PMID 29192011